CLINICAL TRIAL: NCT04562844
Title: Assessment and Rehabilitation of Social Cognition in People With Traumatic Brain Injury
Acronym: CogniSo-TC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A00170-55
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-07

CONDITIONS: Head Injury Trauma; Cognition Disorder
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Intervention Model Description: single group for 1 study and multiples singles cases study for rehabilitation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social cognition (Experimental)
  Interventions: Other: sociale cognition

INTERVENTIONS:
Other: sociale cognition — several social cognition test

SUMMARY:
Patients who have suffered moderate to severe traumatic brain injury (TBI) frequently develop behavioural changes, which can have deleterious consequences on interpersonal relationships, social, family and professional reintegration. They are a source of difficulties (burden) for family and friends. Social cognition covers four functions: recognition of social cues; empathy; attribution of intentions to a third party, or theory of mind; and adjustment of social behaviour according to context. This study has two parts: 1/ Evaluation, using a cognitive approach, of the different components of social cognition after moderate to severe traumatic brain injury, and of its repercussions in daily life and on family and friends.

2/ Creation of a specific re-education method for the different modules of social cognition and study of its effectiveness.

DETAILED DESCRIPTION:
First objective: to study in a systematic way in the same group of TBI patients the different domains of social cognition and the relationships between these different sub-domains in these patients, as well as the relationships between these deficits and the more global cognitive functioning (executive functions), and to evaluate their repercussions in daily life (activity limitations and participation restrictions).

Second objective: to develop and evaluate the effectiveness of a specific rehabilitation protocol for social cognition, adjusted to each profile, according to the disorders of the components of social cognition found in each patient. We make the hypothesis that not all patients will present homogeneous deficits and we also wish to bring elements of knowledge on the sub-domains of social cognition that can be "mobilized" by therapeutic means based on cognitive training adapted to each patient. The methodology envisaged is based on an experimental methodology in single repeated case studies, allowing a fine analysis of the architecture of the altered cognitive processes in a given patient and to adapt the rehabilitation protocol in an individualized way.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of legal age,
* Having suffered a moderate to severe traumatic brain injury (Glasgow Coma Scale score of 3 to 12) at least 6 months after the trauma,
* Returned home at least 3 months ago,
* Having given their informed consent,
* Affiliated to the social security system

Exclusion Criteria:

* Psychiatric history,
* Persistent post-traumatic amnesia,
* Instrumental disorders that interfere with taking tests (aphasia, agnosia, neurovisual disorders),
* Mood disorders not stabilized under treatment,
* Patient refuses to participate in the study,
* Participation in another cognitive rehabiltation protocol,
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-09-24 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
social cognition evaluation | 4 hours
  emotional and sociocognitive measurement by questionnaire
humor and global cognition | 4 hours
  attention measurement and mood evolution by questionnaire
social activity measurement | 1 hour
  activity measurement and social cognition evaluation by questionnaire

SECONDARY OUTCOMES:
environnemental measurement | 20 min
  questionnaire
mood measurement | 30 min
  questionnaire
quality of life questionnaire | 1 hour
  questionnaire

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - SAMSAH-UEROS Arceau Anjou, Angers
  - Raymond Poincaré Hospital, Garches
  - Ueros Ugecam, Garches
  - FAM la vie devant soi, Lomme

IPD SHARING:
Plan to Share IPD: No